CLINICAL TRIAL: NCT05648786
Title: Socializing a Science-Based Digital Therapeutic for Substance Use Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Square2 Systems, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Grabinski, Principal Investigator, Square2 Systems, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R44DA047150 (NIH); 2R44DA047150 (NIH)
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Substance Use Disorders; Substance-Related Disorders
Keywords: Digital therapeutic; Smartphone; Social support; Randomized controlled trial
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard outpatient treatment plus Laddr® (Experimental): Laddr® is a smartphone application integrating science-based, therapeutic processes to address a wide range of behavioral problems in the context of a single mobile platform. Laddr includes tools for activating behavior change, solving problems and overcoming obstacles to effective behavior change; teaching skills and providing guidance on the execution of behavior change; and maintaining the end user's motivation to change. It enables longitudinal assessment of individuals' behavior and health status in naturalistic contexts, offers science-based self-regulation behavior change tools of relevance to an array of populations, and enables ongoing monitoring of health behavior. This study evaluates the effectiveness of new features to Laddr®. These new features are designed to be used with a support person, which could include a friend, family member, or acquaintance.
  In addition to Laddr®, participants will receive standard outpatient substance use disorder treatment.
  Interventions: Behavioral: Laddr® plus Behavioral- Group and individual counseling
- Standard outpatient treatment (Active Comparator): The active control condition consists of standard outpatient treatment for substance use disorders. Outpatient treatment will include a range of services, including group counseling, individual counseling, medication treatment, and other recovery support services.
  Interventions: Behavioral: Behavioral- Group and individual counseling

INTERVENTIONS:
Behavioral: Laddr® plus Behavioral- Group and individual counseling — Smartphone application utilizing the Community Reinforcement Approach (CRA) to facilitate social support in substance use treatment.
  Outpatient treatment will include a range of services, including group counseling, individual counseling, medication treatment, and other recovery support services.
  Arms: Standard outpatient treatment plus Laddr®
Behavioral: Behavioral- Group and individual counseling — The active control condition consists of standard outpatient treatment for substance use disorders. Outpatient treatment will include a range of services, including group counseling, individual counseling, medication treatment, and other recovery support services.
  Arms: Standard outpatient treatment

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an intervention delivered on a smartphone. This study examines whether this intervention might improve treatment outcomes for people with substance use disorders. The intervention, called Laddr®, is a smartphone application ("app") that provides information and skills that can help people stop using substances. The social version of Laddr® being tested in this study has new features that allow people in treatment for substance use disorders to include a support person in their treatment journey, including a friend, family member, or other acquaintance. This research study will compare the effectiveness of Laddr® in combination with standard outpatient substance use treatment to standard treatment only for substance use disorders.

DETAILED DESCRIPTION:
Digital therapeutics, or software used to prevent, treat, or manage a medical disorder or disease, are redefining the future of healthcare by providing on-demand access to state-of-the-science care. Digital therapeutics have been developed to treat a wide range of disorders, including substance use disorders (SUD). Developed by the study Principal Investigator (PI) and Co-Investigator (Co-I), Laddr® is a unique mobile platform integrating science-based therapeutic processes to address a wide range of behavioral problems, including SUD.

The current project expands Laddr® to allow users to engage a support network of their choosing in their journey of behavioral change. Individuals can share data from Laddr about their successes and challenges, and their support network can offer anytime/anywhere social support. Social support will be embedded within a strongly science-based digital therapeutic process - thus providing support persons with a clear framework in which to offer support. Research has shown that engaging a support network of non-substance users (e.g., family members, friends) in one's SUD treatment can greatly enhance treatment outcomes - and is aligned with the "community reinforcement" tenet of the CRA treatment model. Interventions that leverage social support networks can help keep individuals engaged in treatment, reinforce their successes, and help them troubleshoot challenges.

This pragmatic, randomized controlled trial aims to evaluate the effectiveness of the social version of Laddr® in improving SUD treatment outcomes. Adults entering outpatient SUD treatment at the Farnum Center in Manchester, New Hampshire (NH) will be offered the opportunity to be randomized to 12 weeks of standard treatment (treatment as usual [TAU] arm), or standard treatment plus the social version of Laddr® (Laddr® arm). The primary study outcome is retention in SUD treatment (time to treatment dropout), and the investigators hypothesize that participants receiving Laddr® will be retained in treatment for a longer duration. Secondary outcomes include participant substance use (self-report and urine toxicology), stages of change, coping skills, recovery capital, and treatment acceptability.

ELIGIBILITY:
Inclusion Criteria:

* In first 30 days of new outpatient treatment episode at the Farnum Center
* 18 years of age or older
* Ability to provide informed consent
* Has access to a functioning smartphone
* Able to identify a support person who can participate in the study with them
* Available to participate for the full duration of the study.

Exclusion Criteria:

* Inability to understand or read English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Retention in treatment Retention in treatment Retention in treatment Retention in treatment Retention in treatment | 16 weeks
  Time between randomization and dropout from standard outpatient treatment

SECONDARY OUTCOMES:
Substance use composite measure (Timeline Follow-Back and Urine Toxicology) | 16 weeks
  Abstinence from substance use. Each half-week of treatment will be categorized as abstinent if the toxicology screen is negative and the self-report indicates no drug use/heavy drinking days. If self-report is missing but the urine screen is positive, the half-week will be scored as not abstinent.
Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) | 16 weeks
  Motivation to change substance use. SOCRATES scores are calculated for three domains of change readiness, Recognition (Range: 7-35), Ambivalence (Range: 4-20), and Taking Steps (Range: 8-40), with higher scores indicating higher levels of change readiness.
Coping Strategies Scale (CSS) | 16 weeks
  Assessment of strategies to refuse drugs, solve problems, avoid high risk situations, cope with cravings, manage emotions, and develop assertiveness. The CSS total score is calculated by taking the mean of all items and will range from 1-4 points, with higher scores indicating more frequent use of coping strategies.
Assessment of Recovery Capital (ARC) | 16 weeks
  Assessment of resources to help in recovery. This 50 item assessment is scored by assigning one point for each "Yes" response. Total scores range from 0-50 with higher scores indicating higher recovery capital.
Treatment acceptability | 16 weeks
  Acceptability of the treatment model will be assessed among both patients in SUD treatment (for both treatment conditions) and support persons in the Laddr condition. Acceptability will be comprised of both utility and satisfaction with each treatment model across five indicators (0-10 point scales) asking how useful (not at all to very), how much new information (none to a great deal), how easy to understand (very easy to very difficult; reverse coded), how interesting (not at all to very), and how satisfied (not at all to very) they were with the treatment condition to which they were exposed.

CONTACTS AND LOCATIONS:
Locations (1):
- Farnum Center, Manchester, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No